CLINICAL TRIAL: NCT03244696
Title: Behavior and Activity Monitoring in Multiple Sclerosis
Brief Title: Behavior and Activity Monitoring in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Ruchika Prakash, Ruchika Prakash, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014H0483
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Sclerosis; Demyelinating Autoimmune Diseases, Central Nervous System; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases; Immune System Diseases; Physical Activity; Walking; Hydration; Lifestyle Intervention; Health Behavior Tracking; Inflammatory Biomarkers; Neurodegenerative Disease
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Sclerosis; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases; Immune System Diseases; Motor Activity; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step Tracking (Experimental): Participants will track their physical activity in steps using an accelerometer for a period of 6 months. Participants will monitor their overall step-count using the accelerometer, and daily and weekly summaries of their progress provided by the experimenters.
  Interventions: Behavioral: Step Tracking
- Water Tracking (Active Comparator): Participants will track their water-intake using a smart water bottle for a period of 6 months. Participants will monitor their overall water consumption using a smart water bottle, and daily and weekly summaries of their progress provided by the experimenters.
  Interventions: Behavioral: Water Tracking

INTERVENTIONS:
Behavioral: Step Tracking — The step tracking intervention is designed to increase physical activity through the use of self-monitoring and brief motivational materials. The motivational materials will be delivered at various points during the intervention. Participants are not required to access and read these materials, however, the hope is these materials will aid in study and goal adherence. Engagement in the intervention will be tracked by the experimenters using the behavioral data gathered by the tracker.
  Arms: Step Tracking
Behavioral: Water Tracking — The water tracking intervention is designed to increase water intake, to a healthy level, through the use of self-monitoring and brief motivational materials.The motivational materials will be delivered at various points during the intervention. Participants are not required to access and read these materials, however, the hope is these materials will aid in study and goal adherence. Engagement in the intervention will be tracked by the experimenters using the behavioral data gathered by the tracker.
  Arms: Water Tracking

SUMMARY:
The investigators propose to conduct a randomized 6-month intervention study comparing cognitive functioning in individuals with relapsing-remitting multiple sclerosis assigned to either a physical activity or an active water-intake control group. Individuals will complete pre-, mid- and post-assessments of cognitive, physical, and behavioral functioning.

DETAILED DESCRIPTION:
Interventions to increase physical activity through aerobic exercise are some of the only known treatment options to improve domains of cognition such as executive function. While increased physical activity is associated with preserved cortical functioning during exogenous executive functioning tasks in older adults, little is known about the relationship between physical activity and executive functioning in multiple sclerosis. Thus, the investigators propose to conduct a randomized 6-month accelerometry-based intervention designed to increase overall physical activity in sedentary relapsing-remitting multiple sclerosis with known cognitive challenges. The overall objective is to determine how a 6-month activity tracking intervention impacts the behavioral, neural and mechanistic associations between physical activity and cognitive functioning. All individuals who contact the Clinical Neuroscience Laboratory (CNL) with interest in this study will undergo a phone/online screening assessing inclusion/exclusion criteria. Those participants meeting I/E criteria will be invited to the lab for 2 pre-assessment sessions, one session at midpoint, and 2 post-assessment sessions at the completion of the 6 month intervention. Participants will also be asked to complete a number of online questionnaires following the first assessment session. The two pre-assessments will involve a through measure of cognitive functioning, both through the use of neuropsychological batteries and neuroimaging, and inflammatory markers through collection of a blood sample. Following the pre-assessment sessions, conducted by blind personnel, participants will be randomized to one of the two groups. Participants will be asked to self-monitor their assigned health behavior with the aid of a behavioral tracker (accelerometer or smart water bottle). Via a mobile application designed by the laboratory, participants will receive daily and weekly summaries of their health behavior progress, and motivational materials to encourage goal attainment. The 6-month intervention will involve minimal contact from study coordinators. Participants who do not adhere to study goals will be contacted by a study coordinator via phone who will use motivational interviewing to promote behavior change. Following the 6-month intervention the 2 assessment sessions will be repeated to obtain post-intervention data for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite diagnosis of Relapsing-Remitting Multiple Sclerosis
* Score higher than 23 on the Mini-Mental Status Examination (MMSE)
* Expanded Disability Status Scale (EDSS) under 5.5
* Right-handed

Exclusion Criteria:

* Clinically isolated syndrome or progressive MS subtype
* Presence of any other neurological disorders
* Presence of psychiatric disorder diagnosed by a licensed mental health provider in the last two years
* Clinically definite relapse or use of high dose corticosteroids within the last 30 days
* Recreational drug use in the last 6 months
* Without access to a smart phone or no access to the internet
* Current use of accelerometer, pedometer, and/or physical activity monitoring equipment
* Presence of ferromagnetic implanted devices or self-reported claustrophobia

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Performance on a Latent Measure of Working Memory/Processing Speed | Baseline, 3 months, and 6 months
  Change in a latent factor of working memory/processing speed will be examined from pre to post intervention. This latent factor will be created using baseline performance on measures from the Minimal Assessment of Cognitive Functioning in Multiple Sclerosis battery (MACFIMS), the NIH Toolbox Cognition Battery (NIHTB-CB), and the processing speed and working memory measures from the Wechsler Adult Intelligence Scale (WAIS-IV) before, during (at midpoint), and after the intervention. Higher scores on this factor represent better working memory/processing speed performance. Investigators hypothesize changes in cognitive performance, specifically in the domains of working memory and processing speed.

SECONDARY OUTCOMES:
Changes in the Functional Architecture of the MS Brain during Working Memory | Baseline and 6 months
  Before and after the intervention, participants will undergo a brain imaging scan using functional Magnetic Resonance Imaging (fMRI) technology. Network strength in the working memory connectome during the NBack task will be the primary fMRI-based neuroimaging measure. Higher network strength in the working memory connectome represent greater connections between brain edges associated with high working memory performance. Participants in the physical activity group will show increased network strength in a connectome-based model of working memory performance.
Changes in the Functional Architecture of the MS Brain during Processing Speed | Baseline and 6 months
  Before and after the intervention, participants will undergo a brain imaging scan using functional Magnetic Resonance Imaging (fMRI) technology. Network strength in the processing speed neuromaker during the Symbol Digit Modalities Test will be the outcome variable. Higher network strength in the processing speed neuromarker represent greater connections between brain edges associated with high processing speed performance. Participants in the physical activity group will show increased network strength in this neuromarker of processing speed.
Changes on a Self-Report Measure of Depression | Baseline, 3 months, and 6 months
  Participants will be administered Beck Depression Inventory-II before, at mid-point, and after the intervention. This measure assesses self-reported depressive symptoms with a range of 0-63 with higher scores characterizing higher endorsement of depressive symptoms. Changes in scores will indicate effects of the intervention on symptoms of depression.
Changes on a Self-Report Measure of Anxiety | Baseline, 3 months and 6 months
  Participants will be administered the Penn State Worry Questionnaire before, at mid-point and after the intervention. This measure assesses self-reported worry symptoms with a range of 16-80. High scores on this measure represent higher levels of chronic worrying. Change on this measure will be assessed to determine the impact of the intervention on symptoms of worry.
Changes on a Self-Report Measure of Perceived Stress | Baseline, 3 months and 6 months
  Participants will be administered the Perceived Stress Scale before, at mid-point and after the intervention. This measure assesses perceived stress with a range of 0-40. High scores on the perceived stress scale represent higher levels of stress. Change on this measure will indicate impact of the intervention on symptoms of stress.
Changes on a Self-Report Measure of Quality of Life | Baseline, 3 months and 6 months
  Participants will be administered the Satisfaction with Life Scale and the World Health Organization Quality of Life Scale before, at mid-point, and after the intervention. Standardized scores for the two measures will be merged to create a composite score for quality of life. High scores on this composite measure would represent higher quality of life. Differences in the composite score of quality of life will reveal changes in quality of life as a function of the intervention.
Changes on a Self-Report Measure of Sleep Quality | Baseline, 3 months and 6 months
  Participants will be administered the Pittsburgh Sleep Quality Index before, at mid-point, and after the intervention. This measure assesses sleep quality with a range of 0-21. Higher score on this measure represents greater difficulty with sleep. Score changes on this measure will indicate changes in sleep quality as a function of the intervention.
Changes on a Self-Report Measure of Fatigue | Baseline, 3 months and 6 months
  Participants will be administered the Modified Fatigue Impact Scale before, at mid-point and after the intervention. This measure assesses self-reported fatigue with a range of 0-84. High scores on this measure represent higher levels of experienced fatigue. Differences in scores on this measure will indicate changes in fatigue as a function of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchika S Prakash, PhD, Principal Investigator — Ohio State University
Locations (1):
- Department of Psychology, The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phansikar M, Duraney EJ, Manglani HR, Shankar A, Roberts C, Andridge R, Nicholas JA, Petosa R, Prakash RS. TRACking health behavior in people with multiple sclerosis: Effects of a randomized trial on physical activity and working memory. Rehabil Psychol. 2025 Aug;70(3):227-239. doi: 10.1037/rep0000578. Epub 2024 Aug 29. PMID 39207422
- [Derived] Manglani HR, Phansikar M, Duraney EJ, McKenna MR, Canter R, Nicholas JA, Andridge R, Prakash RS. Accelerometry measures of physical activity and sedentary behavior: Associations with cognitive functioning in MS. Mult Scler Relat Disord. 2023 Nov;79:104963. doi: 10.1016/j.msard.2023.104963. Epub 2023 Aug 28. PMID 37690438
- [Derived] Manglani HR, Fountain-Zaragoza S, Shankar A, Nicholas JA, Prakash RS. Employing Connectome-Based Models to Predict Working Memory in Multiple Sclerosis. Brain Connect. 2022 Aug;12(6):502-514. doi: 10.1089/brain.2021.0037. Epub 2021 Sep 28. PMID 34309408